CLINICAL TRIAL: NCT00728143
Title: Therapeutic Trials of Low Glycemic Index Foods and Dietary Fiber in the Management of Diabetes, Hyperlipidemia and Renal Disease
Brief Title: Blood Glucose Response to Highly Viscous Polysaccharide Enriched Biscuits in Healthy and Diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Director of Research, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1_Jenkins
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Healthy subjects
  Interventions: Dietary Supplement: Highly viscous polysaccharide enriched biscuits
- 2 (Experimental): Diabetic subjects
  Interventions: Dietary Supplement: Highly viscous polysaccharide enriched biscuits

INTERVENTIONS:
Dietary Supplement: Highly viscous polysaccharide enriched biscuits — 10 g of highly viscous polysaccharide
  Other Names: HVP

SUMMARY:
Our objective was to test whether the highly viscous polysaccharide incorporated into the biscuit formulation would reduce the postprandial blood glucose response equally in healthy subjects and individuals with type 2 diabetes.

DETAILED DESCRIPTION:
Despite significant achievements in treatment modalities and preventive measures, diabetes has been increasing exponentially. Reduction in both fasting and prolonged postprandial glycemia is of paramount importance in the disease prevention and the delay of diabetic complications. Blood glucose concentration can be reduced by dietary means, and may be influenced by factors such as type and amount of carbohydrate, nature of starch, quantity of protein and fat, dietary fiber content, method of food processing, particle size and food form. Glycemic index (GI) is a measure of the blood glucose-raising ability of the available carbohydrate in foods. Although evidence is often insufficient and individual differences occur, prospective studies and clinical trials have shown that low-GI diets may reduce the risk of diabetes and improve glycemic control in diabetes.

High postprandial plasma glucose level can increase severity of diabetes and foods which raise the blood glucose level least for a given carbohydrate content are most suitable for individuals with type 2 diabetes. Lower postprandial glycemia is also important for healthy subjects to prevent diabetes.

High fiber diets have been recommended for the general population and for the nutritional management of patients with type 2 diabetes. Soluble dietary fiber retards digestion and absorption of the associated dietary carbohydrate, thus flattening the postprandial rise in plasma glucose and insulin concentrations. Some foods such as beta-glucan fiber containing oats and barley, and soluble fibers isolates such as pectin, guar, psyllium, or glucomannan have a high viscosity which gives them the greatest blood glucose lowering effect. Viscous fibers, as a result of their rheological properties, form gel with the food and human digesta and consequently reduce postprandial increases in plasma glucose concentrations in both normal and diabetic subjects in positive relation to their level of viscosity. Insoluble fibers such as cellulose and wheat bran have little effect.

The highly viscous polysaccharide (HVP) added to the study biscuit formulation is a blend of highly viscous soluble fibers (polysaccharides) that act synergistically to develop a higher level of viscosity than any other known dietary fiber in nature. One of the main components of the HVP is glucomannan, a glucose-mannose polysaccharide obtained from grinding the tuber root of Amorphophallus Konjac C. Koch, a plant that has been used as food and remedy for thousands of years in the Far East. Highly refined glucomannan is 3 times more viscous than guar and approximately 7 times more viscous than psyllium. The viscosity of the HVP is amplified further with a viscosity 3-5 times higher than glucomannan alone used in formulation, that is considered to be the highest viscosity single dietary fiber. Previously we and others have shown that the higher viscosity in vitro directly corresponded to lower blood glucose.

ELIGIBILITY:
Inclusion Criteria (arm 1):

* males or non-pregnant females aged 18-75 years and in good health;
* BMI <30 kg/m2.

Exclusion Criteria (arm 1):

* known history of hepatitis, diabetes or a heart condition;
* using medications or fiber supplements;
* any health condition which might affect the results;
* non-compliance with the experimental procedures.

Inclusion Criteria (arm 2):

* documented type 2 diabetes for at least 6 month duration without clinically manifest complications;
* age 18-75 years;
* BMI <30 kg/m2.

Exclusion Criteria (arm 2):

* liver or kidney disease;
* gastrointestinal problems;
* using fiber supplements;
* non-compliance with the experimental procedures;
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1989-08; Primary Completion 1989-11 (Actual); Study Completion 1989-11 (Actual)

PRIMARY OUTCOMES:
Glycemic Index | Two months

SECONDARY OUTCOMES:
Palatability | Two months

CONTACTS AND LOCATIONS:
Overall Officials: David Jenkins, MD, PhD, DSc, Principal Investigator — Unity Health Toronto

REFERENCES:
- [Derived] Jovanovski E, Jenkins A, Dias AG, Peeva V, Sievenpiper J, Arnason JT, Rahelic D, Josse RG, Vuksan V. Effects of Korean red ginseng (Panax ginseng C.A. Mayer) and its isolated ginsenosides and polysaccharides on arterial stiffness in healthy individuals. Am J Hypertens. 2010 May;23(5):469-72. doi: 10.1038/ajh.2010.5. Epub 2010 Feb 4. PMID 20134405